CLINICAL TRIAL: NCT00928200
Title: Intravenous Erwinase for Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia and Allergy to E. Coli Asparaginase (IND 104224)
Brief Title: Erwinase for Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) (IND 104224)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was terminated due to lack of accrual.
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2006-002
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Results first posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2018-07

CONDITIONS: Relapsed Acute Lymphoblastic Leukemia; Allergy to PEG e.Coli Asparaginase; Allergy to Native e.Coli Asparaginase
Keywords: Relapsed; Allergy; Erwinia; Acute; Lymphoblastic; Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence; Hypersensitivity; Leukemia | interventions — Asparaginase; asparaginase erwinia chrysanthemi recombinant; Vincristine; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate; Doxorubicin; Cytarabine; Methotrexate; Dexrazoxane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients receive Vincristine, Dexamethasone, Doxorubicin, and Cytarabine. Dexrazoxane optional on Day 1. Erwinase is started between Days 3-5 and is given every M-W-F for a total of 10 doses. Patients with CNS 1 or 2 receive Methotrexate intrathecally on Day 15. Patients with CNS 3 receive Triple Intrathecal Therapy (Methotrexate, Cytarabine and Hydrocortisone) on Days 8, 15, and 22.
  Interventions: Drug: Erwinase; Drug: Vincristine; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Cytarabine; Drug: Methotrexate; Drug: Triple Intrathecal Therapy; Drug: Dexrazoxane

INTERVENTIONS:
Drug: Erwinase — The dose of Erwinase will be assigned at study entry. The first dose of Erwinase wil be given between Days 3-5 and will continue on a M-W-F schedule for a total of 10 doses.
  Erwinase will be administered as a 2-hour intravenous infusion.
  Other Names: Asparaginase; Elspar; Kidrolase; L-Asparaginase; Erwinia L-Asparaginase
Drug: Vincristine — 1.5 mg/m2/dose IV push (maximum single dose 2 mg) on Days 1, 8, 15 and 22
  Other Names: Oncovin; Vincasar Pfs; Vincristine Sulfate; LCR; VCR
Drug: Dexamethasone — 10 mg/m2/day divided BID. Give by mouth days 1-14.
  Other Names: Decadron; Dexasone; Diodex; Hexadrol; Maxidex; Dexamethasone sodium phosphate; Dexamethasone acetate
Drug: Doxorubicin — 60 mg/m2/day IV over 15 minutes on day 1
  Other Names: Adriamycin; Rubex
Drug: Cytarabine — Given Intrathecally at the dose defined by age on day 1. 30 mg for age 1-1.99 50 mg for age 2-2.99 70 mg for age 3 and older
  Other Names: Cytosar-U; Ara-C; Arabinosylcytosine
Drug: Methotrexate — Given Intrathecally to all patients who are CNS 1 or 2 at study entry. Dose defined by age. Given on day 15 8mg for age 1-1.99 10 mg for age 2-2.99 12 mg for age 3-8.99 15 mg for age 9 and older
  Other Names: Otrexup; Rasuvo; Rheumatrex; Trexall; Amethopterin; Methotrexate Sodium; MTX
Drug: Triple Intrathecal Therapy — Methotrexate, Cytarabine and Hydrocortisone given Intrathecally on day 8, 15 and 22 for patients who are CNS 3 at study entry. Doses determined by age.
Drug: Dexrazoxane — Due to the limited availability of Dexrazoxane (Zinecard®), treatment will be at the discretion of the treating physician. Dose should be 600 mg/m2 as a IV push immediately prior to anthracycline dose (the elapsed time from the beginning of the dexrazoxane dose to the end of the anthracycline infusion should be 30 minutes or less).
  Other Names: Zinecard

SUMMARY:
This is a phase I study using the Erwinia form of asparaginase in place of the E. coli form using a standard re-induction regimen (Vincristine, Dexamethasone, Doxorubicin) for patients with relapsed ALL who have developed an allergy to the E. coli formulation. This study will administer the drug intravenously instead of the usual intramuscular route. The dose of Erwinia will be escalated in the absence of dose limiting toxicity. Patients must have first or second relapse ALL with a history of prior systemic reaction to E. coli asparaginase.

DETAILED DESCRIPTION:
Significance

1. Substitution of Erwinase after E.coli asparaginase allergy has been standard practice despite the paucity of evidence regarding its efficacy and uncertainty about dose. Definition of an appropriate dose and schedule of Erwinase that provides reliable asparagine depletion may be useful for patients with clinical allergy to E. coli asparaginase, both in first remission or after relapse.
2. Patients in relapse may have a different level of asparagine synthesis than patients maintaining remission and require different asparaginase dosing.5
3. Intravenous administration provides more rapid and predictable asparagine depletion with less discomfort and danger of bleeding for often thrombocytopenic patients than intramuscular administration.
4. Vincristine, doxorubicin, asparaginase, and dexamethasone with dexrazoxane is clinically relevant for a population with first marrow relapse.
5. Vincristine, doxorubicin, asparaginase, and dexamethasone with dexrazoxane is clinically relevant for a population with second marrow relapse, if the duration of CR2 > 18 months year.

ELIGIBILITY:
Inclusion Criteria The eligibility criteria listed below are interpreted literally and cannot be waived.

1. Age Patients must be >1 and < 21 years of age when enrolled onto this study.
2. Diagnosis Patients must have relapsed or refractory ALL with a M3 marrow (marrow blasts >25%) who have had no more than two prior therapeutic attempts. Patients with CNS 1, 2, or 3 or testicular disease are eligible. (See section 11.3 for CNS definitions)
3. E. coli Asparaginase Allergy Patients must have a history of prior systemic allergic reaction to E. coli asparaginase (native or pegylated), such as urticaria, wheezing, or anaphylaxis. Local reactions are not sufficient.
4. Performance Level Karnofsky > 50% for patients > 10 years of age and Lansky > 50% for patients < 10 years of age.
5. Prior Therapy Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.

   1. Patients may be in first or second relapse and should not have received more than 2 induction attempts (including frontline therapy).
   2. Prior anthracycline exposure: Patients must have less than 400mg/m2 lifetime exposure of anthracycline chemotherapy.
   3. Stem Cell Transplant (SCT): Patients are eligible after allogeneic stem cell transplant as long as patients are not actively being treated for graft-versus-host-disease (GvHD).
   4. Patients may have received previous therapy using intramuscular (IM) Erwinase. Patients who have received Erwinase intravenously will be excluded.
6. Reproductive Function

   1. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

Exclusion Criteria

1. Prior Stroke Patients with a prior history of asparaginase associated stroke are excluded. Patients with a history of other asparaginase related deep-venous thromboses (including intra-cranial thromboses without evidence of stroke or hemorrhage) are eligible.
2. Down Syndrome Patients with Down Syndrome will be excluded.
3. Prior Pancreatitis Patients with prior history of Grade 2 or greater asparaginase-induced symptomatic pancreatitis will be excluded.
4. Renal Function Patients will be excluded if their serum creatinine is > 1.5 x the upper limit of normal for age at the institution's laboratory.
5. Liver/Pancreatic Function

   Patients will be excluded if their lab results are as follows:
   1. Direct bilirubin > 1.5x the institutional ULN for age. A total bilirubin result that is less than 1.5 times the institutional ULN for age may be used for eligibility if a direct bilirubin result is not available.
   2. SGPT (ALT) > 4 x institutional ULN
   3. Amylase or Lipase > 2 x institutional ULN
6. Cardiac Function Patients will be excluded if their shortening fraction by echocardiogram is less than the institutional normal for age or an ejection fraction by MUGA is less than the institutional normal for age.
7. Infection Patients will be excluded if they have an active uncontrolled infection.
8. Patients planning on receiving other investigational agents while on this study. (An investigational agent is defined as any drug not currently approved for use in humans.)
9. Patients planning on receiving other anti-cancer therapies while on this study.
10. Patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
11. Patients who have started protocol therapy prior to enrollment. Patient may still enroll if IT therapy was given within 72 hours of study enrollment as part of the diagnostic lumbar procedure.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2009-04-13; Primary Completion 2010-06-04 (Actual); Study Completion 2010-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Grossman, MD, Study Chair — Children's Hopital New York; Paul Gaynon, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: All patients receive Vincristine, Dexamethasone, Doxorubicin, and Cytarabine. Dexrazoxane optional on Day 1. Erwinase is started between Days 3-5 and is given every M-W-F for a total of 10 doses. Patients with CNS 1 or 2 receive Methotrexate intrathecally on Day 15. Patients with CNS 3 receive Triple Intrathecal Therapy (Methotrexate, Cytarabine and Hydrocortisone) on Days 8, 15, and 22.
  Erwinase: The dose of Erwinase will be assigned at study entry. The first dose of Erwinase wil be given between Days 3-5 and will continue on a M-W-F schedule for a total of 10 doses.
  Erwinase will be administered as a 2-hour intravenous infusion.
  Vincristine: 1.5 mg/m2/dose IV push (maximum single dose 2 mg) on Days 1, 8, 15 and 22
  Dexamethasone: 10 mg/m2/day divided BID. Give by mouth days 1-14.
  Doxorubicin: 60 mg/m2/day IV over 15 minutes on day 1
  Cytarabine: Given Intrathecally at the dose defined by age on day 1. 30 mg for age 1-1.99 50 mg for age 2-2.99 70 mg for age 3
Period: Overall Study
Arm/Group | Single Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of a Dose-Limiting Toxicity
Description: The MTD in each stratum will be the highest dose at which 1 or fewer of six patients experience DLT during cycle 1 of therapy.
Time Frame: Beginning with the first dose of investigational product until 30 days following the last dose of Erwinase
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Response Rate and Minimum Residual Disease
Description: Disease response evaluated by examination and labs. MRD evaluated from marrow samples.
Time Frame: After completion of treatment course
Population: Study closed early due to lack of accrual, and insufficient data were collected for performing this analysis.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

3. Secondary Outcome: Asparaginase Activity
Description: Activity levels assessed from PK sampling
Time Frame: PK samples to be collected Pre-Tx, and and Erwinase Doses 3, 6 and 9 and Day 29
Population: Study closed early due to lack of accrual and insufficient data were collected to perform this analysis.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The definition of AE and SAE do not differ from the clinicaltrials.gov definitions.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=1)
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=1)
Agitation (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood fibrinogen (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Injection site reaction NOS (Injury, poisoning and procedural complications) | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 1
Neutrophil count (Blood and lymphatic system disorders) | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Vomiting NOS (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study closed early due to lack of accrual and insufficient funding. Only one patient was enrolled. This patient completed the protocol therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days